CLINICAL TRIAL: NCT06872151
Title: Evaluation of the Effectiveness of a Gel Containing a Propionibacterium Extract in Wound Healing and Symptom Relief, Such as Pain, Itching, and Burning, in the Postoperative Period of Open Excisional Hemorrhoidectomy
Brief Title: Evaluation of the Effectiveness of a Topical Medical Device in Wound Healing and Symptom Relief in the Postoperative Period of Open Excisional Hemorrhoidectomy (The Emor Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Policlinico Umberto I (Other); Hospital San Pietro Fatebenefratelli (Other); University Hospital of Ferrara (Other); ASL Roma 6 (Other)
Responsible Party: Principal Investigator, Simona Deidda, Assistant professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TheHemorrStudy_Vers_05_02_2024
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-03

CONDITIONS: Anus Diseases; Gastrointestinal Diseases; Intestinal Diseases; Cicatrization; Hemorrhoids; Hemorrhoids Third Degree
Keywords: hemorrhoids; epithelialization; Anal diseases; hemorrhoidectomy
MeSH Terms: conditions — Anus Diseases; Gastrointestinal Diseases; Intestinal Diseases; Cicatrix; Hemorrhoids | interventions — Hyaluronic Acid; Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gel containing a Propionibacterium extract (Experimental)
  Interventions: Device: Gel containing a Propionibacterium extract
- Hyaluronic acid and silver sulfadiazine (Active Comparator)
  Interventions: Drug: Hyaluronic acid and silver sulfadiazine

INTERVENTIONS:
Device: Gel containing a Propionibacterium extract — Patients will apply 1 ml of gel (equal to one phalanx) twice a day for 20 days, manually at the anal level and in the perianal area. In the morning, after defecation and in the evening before going to bed.
  Arms: Gel containing a Propionibacterium extract
Drug: Hyaluronic acid and silver sulfadiazine — Patients will apply 1ml of gel (equal to a phalanx) twice a day for 20 days, manually at the anal level and in the perianal area. In the morning, after defecation and in the evening before going to bed.
  Arms: Hyaluronic acid and silver sulfadiazine

SUMMARY:
This multicenter randomized controlled phase IV trial aims to compare the clinical efficacy of a gel containing a Propionibacterium extract and a gel with hyaluronic acid and silver sulfadiazine in the degree of epithelialization of post-operative wounds of open excisional hemorrhoidectomy.

The main questions it aims to answer are:

* To compare the efficacy of the two medical devices in the degree of epithelialization in the postoperative period of open excisional hemorrhoidectomy, at 0, 10, 20 and 40 days from the beginning of treatment.
* To evaluate the effectiveness of these devices in alleviating: pain, itching, burning, and the type of bowel habit Participants will be randomized, at the beginning of the study, to one of the two treatments, and the efficacy of the two medical devices will be evaluated at 0, 10, 20 and 40 days from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Open excisional hemorrhoidectomy, with removal of at least 3 groups
* Age between 18 and 75 years

Exclusion Criteria:

* Patients who do not consent to the study
* Opioid-dependent patients, chronic use of analgesics
* Fecal incontinence
* Anorectal neoplasms
* Immunosuppressive treatments (e.g., chemotherapy, radiotherapy, etc.)
* Chronic inflammatory bowel diseases
* Pregnancy
* Patients with major psychiatric disorders
* Known allergy to the components of the treatments under study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Degree of epithelialization | From baseline to visit 3 (40 days after the start of the treatment)
  The degree of epithelialization of the fissure was determined at each visit and stratified using 3 levels (1 to 3) corresponding to:
  1. < 50%
  2. > 50%
  3. 100% (complete healing)

SECONDARY OUTCOMES:
Burning and pain | From baseline to visit 3 (40 days after the start of the treatment)
  Visual analogue scale (VAS) (minimum score = 0, maximum score = 10)
Itching | From baseline to visit 3 (40 days after the start of the treatment)
  Visual analogue scale (VAS) (minimum score = 0, maximum score = 10)
Bowel movements | At visit 3 (40 days after the start of the treatment)
  Bristol Scale (minimum score =1, maximum score =7)

CONTACTS AND LOCATIONS:
Overall Officials: Deidda, Principal Investigator — University of Cagliari
Locations (1):
- Policlinico Universitario Monserrato "Duilio Casula" - AOU Cagliari, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No